CLINICAL TRIAL: NCT06679868
Title: Role of ALBI Score and Sarcopenia As Prognostic Predictors Among Hospitalized Cirrhotic Patients with Hepatic Encephalopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Saad Ahmed Abu Elsoud, HSAAD, Assiut University
Other Study IDs: ALBI and Sarcopenia in LC
Record Dates: First submitted 2024-09-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate the role of ALBI score in predicting prognosis and hospital mortality of hospitalized cirrhotic patients with hepatic encephalopathy.

To verify the best scoring system for predicting prognosis and survival among those patients.

To investigate whether the presence of sarcopenia could add to the prognostic role of ALBI score.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a brain dysfunction caused by impaired liver functions and/or portosystemic shunting. It is one of the most serious complications of liver cirrhosis that leads to a signifcantly impaired quality of life and frequent hospitalizations.

Although the pathogenesis of HE is complex ,accumulation of ammonia ,systemic inflammation, and oxidative stress play a pivotal role .Multiple organs are involved in whole body homeostasis of ammonia, with the liver being a key site .As cirrhosis leads to decline in capacity of liver to detoxify ammonia, skeletal muscle plays a compensatory in ammonia metabolism and clearance .Liver function largely reflect prognosis of liver disease,The ALBI score was originally developed as a measure of liver function in patients with HE.It was developed by putting all of the original components of the Child-Pugh (CTP) score into a multivariable model, the clinical features, (Ascites, Encephalopathy and INR) ,were shown to be redundant in that the entire prognostic value of the CTP score could be explained by just albumin and bilirubin levels in an appropriate formulation derived from multivariable model.As with the CTP and MELD scores, both of which were introduced for specific clinical situation and extended to more general application, the same has happened with ALBI.Increasingly, ALBI score is applied as a preferred measure of liver function due to its objectivity and sensitivity for minor liver function deterioration . In comparison to the MELD score, The ALBI score is sufficiently sensitive of liver function ,thus it might be expected to predict longer-term mortality in patients with cirrhosis, better than the MELD score, which would be expected to predict shorter-term mortality in patients with decompensated cirrhosis or liver failure. A study showed clearly that the ALBI score is the most accurate scoring system in predicting prognosis, followed by CTP, CLIF-SOFA, MELD-Na. Furthermore, it has been shown that the ALBI score is the strongest independent predictor of mortality among other scores. The presence of sarcopenia leads to higher risk of HE. Muscle depletion defined by mid arm circumference is associated with development of covert and overt HE

ELIGIBILITY:
Inclusion Criteria:

* All cirrhotic patients with hepatic encephalopathy admitted to Al-Rajhi liver hospital.

Exclusion Criteria:

* Patients with acute hepatic failure and those with previous portosystemic surgery or TIPS.
* Patients with prior liver or other organs transplantation.
* End stage renal disease(ESRD), and HCC or other solid tumors.
* Patients on marivan for any cause.
* Patients with extra-hepatic biliary obstruction.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
1- Evaluation of the role of ALBI score in predicting prognosis and hospital mortality of hospitalized cirrhotic patients with hepatic encephalopathy. 2- Verification of the best scoring system for predicting prognosis and survival among those patients | ALBI score/at admission and follow up of patients /after 1 month
  ALBI score can be assessed by following formula : 0.66Xlog(bilirubin.mg/dl)_0.085X(albumin.g/dl)The cut-off points for ALBI grades are:Grade I : less than -2.60(lowest mortality risk)Grade II : -2.60 to - 1.39(Intermediate)Grade III : more than -1.39 (Highest ) Follow up of those patients and record of improvement, deterioration or death will be done.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen H, Yang C, Yan S, Liu X, Zhou L, Yuan X. Sarcopenia in cirrhosis: From pathophysiology to interventional therapy. Exp Gerontol. 2024 Oct 15;196:112571. doi: 10.1016/j.exger.2024.112571. Epub 2024 Sep 9. PMID 39236869
- [Background] Hsieh YC, Lee KC, Wang YW, Yang YY, Hou MC, Huo TI, Lin HC. Correlation and prognostic accuracy between noninvasive liver fibrosismarkers and portal pressure in cirrhosis: Role of ALBI score. PLoS One. 2018 Dec 12;13(12):e0208903. doi: 10.1371/journal.pone.0208903. eCollection 2018. PMID 30540824